CLINICAL TRIAL: NCT04174729
Title: System for Quantifying the Functional Strength of the Grip and Pinch Movements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mogi das Cruzes (Other)
Responsible Party: Principal Investigator, Terigi Augusto Scardovelli, Principal Investigator, University of Mogi das Cruzes
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19020219.2.0000.5497
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Hand Injuries and Disorders
MeSH Terms: conditions — Hand Injuries; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hand strength (Experimental): The tests were performed in two sessions lasting 1 hour each. The volunteers used the devices: door handle, tap, door pull handle, switch and door key to quantify hand strength. The tests were performed in two sessions lasting 1 hour each. The volunteers used the devices: door handle, tap, door pull handle, switch and door key to quantify hand strength.
  In the first session, the volunteers performed the movements 3 times in each device of daily living activities with the right limb, with a 1-minute rest interval between the 3 measurements. The entire procedure performed in the session was repeated again after 30 minutes to verify the reliability and reproducibility of the Intra-evaluator test. The Inter-rater test was repeated after 7 days by the second rater to analyze reliability between the rater.
  Interventions: Device: handgrip strength; Device: Door handle device; Device: Tap device; Device: Door pull handle; Device: Linear Switch device; Device: Door Key device

INTERVENTIONS:
Device: handgrip strength — First, the hand measurements of each volunteer were evaluated, followed by the measurement of handgrip strength using the Jamar® dynamometer. And later the tests were performed using the system that contains the 5 devices to quantify the hand strength.
  Other Names: Jamar dynamometer
Device: Door handle device — To evaluate the cylindrical grip movement, a door handle was used, which evaluated the full force in the range of motion.
Device: Tap device — To evaluate the spherical grip movement, a tap was used, which evaluated the full force in the range of motion.
Device: Door pull handle — To assess the hook grip movement, a door pull handle was used, which assessed the full force in the range of motion
Device: Linear Switch device — To evaluate the pulp-pulp pinch movement, a switch was used, which evaluated the full force in the movement of the movement.
Device: Door Key device — To assess the pulp-side pinch movement, a door key was used, which evaluated the full force in the range of motion.

SUMMARY:
This study developed a system to quantify the functional strength of young adults without motor impairment during grip and pinch movement. Making it possible to know the accuracy of the value of these strength, the range of motion performed and whether the grip force was maintained throughout the range of motion. In addition to checking the functionality, reliability and reproducibility of the system.

DETAILED DESCRIPTION:
Quantifying grip and grip movement is essential as it allows for a basis in upper limb functionality. However, when there is access, it causes changes in the hands and changes the motor in relation to the force and range of motion, or generates changes in activities of daily living. Thus, a system with 5 devices, where each one the devices were prints in three-dimensional, and instrumented with force sensor for static-dynamic force analysis e potentiometer for analysis range of motion, during the execution of movements cylindrical grip, spherical grip, hook grip, pulp-pulp pinch, and pulp- side pinch in different activities of daily living. Elaborated a data storage interface through MATLAB® software that allows recording the data of each device. For the system functionality tests, 30 volunteers were selected for both sexes, young adults between 20 and 39 years old, students of the Physiotherapy and Graduate courses of the University of Mogi das Cruzes. The tests are divided into two sessions and are repeated after 7 days of the first test

ELIGIBILITY:
Inclusion Criteria:

* only right-handed individuals,
* male and female,
* have preserved cognitive functions,
* absence of neurological disorder
* who present minimum grip strength by the Jamar ® dynamometer, in the age group of 20-29 years men 45.08 ± 0.67 kg and women of 27.2 ± 0.46 kg, who present minimum grip strength by the dynamometer Jamar ®, aged 30 to 39 years old men 46.05 ± 0.47 kg and women 28.0 ± 0.39 kg, using the mean minus the standard deviation.

Exclusion Criteria:

* Injury to upper limbs such as amputation, recent surgery (6 months), fractures, bruising, pain and musculoskeletal disorders.
* Do not accept to participate in the survey.

Ages: 20 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-10-29 (Actual)

PRIMARY OUTCOMES:
Strength device | 15 minutes
  The strength of the cylindrical grip movement was quantified through the door handle device, the spherical grip strength through the tap device, the hook grip strength through the vertical door pull handle, the pulp-pulp pinch strength through the linear switch device and the pulp-side pinch strength through the key device. The test was quantified 3 times with a 1 minute interval between each test and the force throughout the range of motion.
  Unit of measure: newton (N).

SECONDARY OUTCOMES:
Range of motion in angle | 15 minutes
  The test measured the range of motion of the door handle device, the tap device, door pull handle device and the door key device, 3 times with 1 minute interval for each test, in which all range of motion was measured from its start until its end. Unit of measure: Angle (º).
Range of motion millimeter | 15 minutes
  The test measured the range of motion in a linear switch device 3 times with a 1 minute interval for each test, in which all of the range of motion was measured from its start until its end. Unit measurement: millimeter (mm).

OTHER OUTCOMES:
Anthropometric variables | 5 minutes
  The anthropometric measurement of the right hand was performed using an analog caliper, as it is an important parameter for functional evaluation, as it was of the following anatomical parts: total length of the hand (wrist crease to middle finger tip), longitudinal length of the palm from the hand (wrist crease to the proximal crease of the middle finger) and transverse length of the palm (lateral to medial line of the metacarpophalangeal muscles). Unit of measure: millimeter (mm)
Dynamometer Jamar Strength | 1 minute
  To make the sample more homogeneous, the Jamar ® dynamometer was used to measure grip strength maximum contraction for 3 seconds. A single measurement was performed. Unit of measure: kilogram - force (kgf).

CONTACTS AND LOCATIONS:
Overall Officials: Silvia R Boschi, PhD, Principal Investigator — University of Mogi das Cruzes
Locations (1):
- Silvia Regina Matos da Silva Boschi, Mogi das Cruzes, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No